CLINICAL TRIAL: NCT02539693
Title: Sacrococcygeal Local Anesthesia With Different Doses of Clonidine for Pilonidal Sinus Surgery: A Prospective Randomized Trial
Brief Title: Sacrococcygeal Local Anesthesia With Different Doses of Clonidine for Pilonidal Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 082015
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus | interventions — Clonidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine 75 (Experimental): Patients will receive sacrococcygeal local anesthesia with 75µg/mL of clonidine. The anesthetic mixture will contain: lidocaine 2% 14 mL, bupivacaine 0.5% 5 mL, and clonidine 0.5 mL with 0.5 mL of saline (thus 75 µg/mL).
  Interventions: Drug: Clonidine 75 µg/mL in sacrococcygeal block; Drug: Lidocaine; Procedure: Pilonidal sinus
- Clonidine 150 (Experimental): Patients will receive sacrococcygeal local anesthesia with 150µg/mL of clonidine. The anesthetic mixture will contain: lidocaine 2% 14 mL, bupivacaine 0.5% 5 mL, and clonidine 1 mL (thus 150 µg/mL).
  Interventions: Drug: Clonidine 150 µg/mL in sacrococcygeal block; Drug: Lidocaine; Procedure: Pilonidal sinus

INTERVENTIONS:
Drug: Clonidine 75 µg/mL in sacrococcygeal block — Sacrococcygeal block will be performed using 75 µg/mL clonidine in the anesthetic mixture
  Arms: Clonidine 75
Drug: Clonidine 150 µg/mL in sacrococcygeal block — Sacrococcygeal block will be performed using 150 µg/mL clonidine in the anesthetic mixture
  Arms: Clonidine 150
Drug: Lidocaine — 3 ml lidocaine 1% is injected at each block site
Procedure: Pilonidal sinus — Removal of pilonidal sinus

SUMMARY:
Sacrococcygeal local anesthesia was shown to reduce the time spent in the operating room as well as in the recovery room. In addition, decreased hospital stay and postoperative analgesic consumption.

Given the effectiveness of sacrococcygeal local anesthesia in pilonidal sinus surgery, it would be valuable to study the effect of the local anesthesia with 75µg/mL of clonidine versus 150µg/mL.

DETAILED DESCRIPTION:
Study design and sampling

This is a prospective study with a randomized double-blind design that will be conducted between October 2015 and October 2016.

Patients scheduled for pilonidal sinus surgery will be included. Patients will be randomly distributed to one of 2 groups with 30 patients in each, using the sealed envelope technique. Group one will receive sacrococcygeal local anesthesia with 75µg/mL of clonidine, while group two will receive sacrococcygeal local anesthesia with 150µg/mL of clonidine.

Anesthetic techniques

Being a double-blinded study, a specialized nurse will prepare the syringes for each patient.

Sacrococcygeal local anesthesia technique

The Sacrococcygeal block will be performed with the patient in the prone position. Four injection sites are marked on the skin after aseptic preparation.

The sites are placed as follows: 4 cm below and above the pilonidal sinus and 3 cm lateral to its center on both sides. Therefore a "lozenge" is formed by connecting the 4 sites.

At first, an injection of 0.3 ml lidocaine 1% is injected at each site using an 8-mm 30G needle. Then 4 injections are admitted to each of the 4 injection sites in turn, with equal supply of the anesthetic mixture in the following manner: a 10-mm 27G needle containing the anesthetic mixture is introduced perpendicularly to the skin and the mixture is infiltrated. The needle is partially withdrawn and reinserted at 45 degrees to the skin aiming towards the center of the pilonidal sinus and an injection will be performed. Then the needle is partially withdrawn again and reinserted at an angle of 45 degrees to the skin aiming at one side of the lozenge then at the other side where injections are done.

In case of a multiple pilonidal orifices, a hexagon is done. These sites are then anesthetized as previously described.

Anesthetic mixture

For group 1, the syringe will contain: lidocaine 2% 14 mL, bupivacaine 0.5% 5 mL, and clonidine 0.5 mL with 0.5 mL of saline (thus 75 µg/mL).

As for group 2, the syringes will contain: lidocaine 2% 14 mL, bupivacaine 0.5% 5 mL, and clonidine 1 mL (thus 150 µg/mL).

Depending on each patient's weight and type of pilonidal sinus, the anesthetic mixture might vary from 30 to 40 mL in total.

Data collection

Demographic data, type and duration of surgery will be recorded. Haemodynamics will be registered at all times (pre-operatively, intra-operatively and post-operatively).

Pain will be assessed using VNRS with 0 being no pain and 10 maximum pain for 48 hours post-operatively.

As for postoperative analgesia consumption, patients with a VNRS score less than 3 are given paracetamol 1000 mg each 8 hours. If VNRS is between three and four, patients are given Tramadol Hydrochloride 50-100 mg every 4- 6 hours and if the VNRS score is greater or equal to five, patients receive 1 mg/kg Dolosal.

Return to normal activity will be defined by the ability to sit, walk and work comfortably and will be assessed by calling the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for pilonidal sinus surgery

Exclusion Criteria:

* Patients who have allergic reactions to lidocaine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Compare analgesic consumption using questionnaire | Patients will be followed-up after the operation, an expected average of five days

SECONDARY OUTCOMES:
Time needed to return to normal activity noted by calling the patients | Patients will be followed-up after the operation, an expected average of five days
Pain using verbal numeric rating scale (VNRS) | Patients will be followed-up after the operation, an expected average of five days

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon